CLINICAL TRIAL: NCT01983436
Title: Impact of Manual Lymphatic Drainage on Postoperative Edema of the Face and the Neck After Orthognathic Surgery.Open-label Multicenter Randomized Controlled Trial
Brief Title: Impact of Manual Lymphatic Drainage on Postoperative Edema of the Face and the Neck After Orthognathic Surgery
Acronym: DLMOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PHRIP/12/ADV/DLMOF
Record Dates: First submitted 2013-10-23; First posted 2013-11-14 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Maxillofacial Abnormalities; Post Procedural Discharge
Keywords: Maxillofacial Orthognathic Surgery; Manual lymphatic drainage
MeSH Terms: conditions — Maxillofacial Abnormalities | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual Lymphatic Drainage (Experimental): * 9 daily sessions of manual lymphatic drainage (except on Saturday/Sunday) starting at Day 1 after surgery.
  * 4 more sessions (one every two days).
  Interventions: Other: Manual Lymphatic drainage
- Control (No Intervention): No session of manual lymphatic drainage

INTERVENTIONS:
Other: Manual Lymphatic drainage — Manual lymphatic drainage of the face and the neck is a massage technique that aims to remove an edema of this anatomical region. The technique consists to stimulate the lymph nodes in order to accelerate the lymph flow and to achieve a specific massage to promote the entry of lymph nodes in the initial lymphatics. Massages follow anatomical pathways of vessels and of lymph nodes of the head and the neck. The technique should be smooth and painless.
  Arms: Manual Lymphatic Drainage

SUMMARY:
Orthognathic surgery aims to standardize position of the maxilla and the mandible and therefore chewing, breathing, phonation and swallowing functions. In postoperative, several physical and functional consequences are observed in patients: transient edema of the face, maxillo-mandibular blocking (causing difficulties to eat and occasional weight loss), pain and sensory disturbances (labial or/and chin paresthesias).

Achieving sessions of manual lymphatic drainage by physiotherapist may allow faster decrease of postoperative edema, improved postoperative comfort and mental well-being.

The main objective of this study is to evaluate the efficacy of sessions of manual lymphatic drainage to reduce postoperative edema.

DETAILED DESCRIPTION:
Orthognathic surgery aims to standardize position of the maxilla and the mandible and therefore chewing, breathing, phonation and swallowing functions. In postoperative, several physical and functional consequences are observed in patients: transient edema of the face, maxillo-mandibular blocking (causing difficulties to eat and occasional weight loss), pain and sensory disturbances (labial or/and chin paresthesias).

Achieving sessions of manual lymphatic drainage by physiotherapist may allow faster decrease of postoperative edema, improved postoperative comfort and mental well-being.

The main objective of this study is to evaluate the efficacy of sessions of manual lymphatic drainage to reduce postoperative edema. Secondary objectives of the study are to assess impact of sessions of manual lymphatic drainage on patient comfort (pain, aesthetic discomfort, difficulty in breathing and discomfort in swallowing) and on ental well-being.

Patients allocated to the intervention group will have 13 sessions of manual lymphatic drainage and those allocated in control group will not.

Edema of patients will be measured at day 1, day 8, day 15 and day 22 after surgery by a different physiotherapist than physiotherapist achieving drainage sessions, blind to the randomization group of the patient. At the same time, comfort criteria will be assessed by a visual analogue scale and mental well-being with the General Health Questionnaire (GHQ28).

ELIGIBILITY:
Inclusion Criteria:

* Orthognathic surgery (mandibular osteotomy, maxillary osteotomy or both)
* Providing informed consent.

Exclusion Criteria:

* Postoperative flexible restraint on the chin region.
* Inability to understand and/or follow all scheduled visits.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Assessment of edema using a centimeter scale. | day 22 after surgery
  Assessment in centimeter of the distance between the ear lobes passing under the bottom of the columella, through the chin and passing under the bottom edge of the chin and assessment in centimeter of the neck circumference at 7.5 cm below the lobes ears.

SECONDARY OUTCOMES:
Comfort criteria | Day 22
  Comfort criteria (pain, aesthetic discomfort, difficulty in breathing and discomfort in swallowing) will be assessed by a self-administered questionnaire consisting of visual analogue scale(0-10).
mental well-being. | day 22
  The mental well-being will be assessed by the General Health Questionnaire in its 28 items french version (GHQ-28)

CONTACTS AND LOCATIONS:
Overall Officials: Axel DI VITTORIO, Mr, Principal Investigator — UH TOURS; Julie LEGER, Mrs, Study Chair — UH Tours
Locations (2):
- France (2):
  - UH Montpellier, Montpellier
  - UH Tours, Tours